CLINICAL TRIAL: NCT01269255
Title: A Phase I Trial of Induction Chemotherapy and Chemoradiotherapy With TS-1 and Cisplatin (SP) as First-line Treatment in Patients With High Risk Advanced Gastric Cancer
Brief Title: A Trial of Induction Chemotherapy and Chemoradiotherapy With TS-1 and Cisplatin (SP) as First-line Treatment in Patients With High Risk Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4-2009-0555
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination group (Experimental)
  Interventions: Drug: TS-1 with Cisplatin

INTERVENTIONS:
Drug: TS-1 with Cisplatin — SP CCRT(= TS-1 with Cisplatin concurrent radiation therapy)
  * Step 1: Chemotherapy; TS-1/CDDP #2 cycles
  * Step 2: Chemoradiotherapy; CCRT with weekly TS-1/CDDP
  * Step 3: Surgery therapy

SUMMARY:
A Phase I trial of Induction chemotherapy and Chemoradiotherapy with TS-1 and Cisplatin (SP) as first-line treatment in patients with high risk advanced gastric cancer. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy was effectively used in esophageal cancer, laryngeal cancer and rectal cancer, but gastric cancer are rarely studied in Korea. There is an increasing interest in preoperative radiotherapy in effort to improve survival and increase pathologic complete response in patients with gastric cancer. Chemoradiotherapy may be the best modality in the neoadjuvant setting for high-risk advanced tumors, such as type IV or large type III, N3/bulky N2 metastasis, or locally advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented gastric adenocarcinoma
* Patients must have unresectable disease or high-risk advanced tumor: borrmann type IV, large borrmann type III (>8cm),locally extensive nodal disease (bulky N),locally advanced (T4) tumors,esophageal invasion
* Age: 20 to 75
* ECOG PS: 0 or 1
* Patients with adequate organ function : Absolute neutrophil count > 1.5 x 109 / L, Platelet count > 100 x 109 / L, Hemoglobin > 9 g/dL (by transfusion permitted), Calculated creatinine clearance > 60 ml/min, Serum total bilirubin < 1.5 times upper normal limit (UNL), Serum alanine transaminase (ALT) < 3 times UNL
* Signed informed consent
* Sexually active patients, in conjunction with their partner, must practice birth control during therapy. Female patients in child-bearing age must have negative pregnancy test.
* No other malignancies within the past 5 years except for curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* No prior or concurrent significant medical conditions, including any of the following: Cerebrovascular disease within the past year/ Cardiovascular disease; myocardial infarction within the past year, uncontrolled hypertension while receiving chronic medication, unstable angina, New York Heart Association class II-IV congestive heart failure, serious cardiac arrhythmia requiring medication/ Major trauma, major surgery or open biopsy within the 28 days Serious nonhealing wound, ulcer, or bone fracture/ Evidence of bleeding diathesis or coagulopathy/ Recent history of any active gastrointestinal inflammatory condition
* No lack of physical integrity of the upper GI tract, malabsorption syndrome, or inability to take oral medication
* No bleeding from primary tumor or gastrointestinal stenosis
* sufficient oral intake
* No prior surgery for gastric cancer except for endoscopic membrane resection (EMR)
* No known peripheral neuropathy ≥ 1
* No prior chemotherapy
* No prior radiotherapy

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Metastasis to the sites out of abdomen (liver or other hematogenous metastasis)
* Patients with definite ascites in pre-operative abdomen CT
* documented inoperable peritoneal seeding disease determined by exploratory laparotomy
* Past or concurrent history of neoplasm other than gastric cancer, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions: History of significant neurologic or psychiatric disorders including dementia or seizures/ Active uncontrolled infection/ Severe hypercalcemia of above 12 mg/dL uncontrolled with bisphosphonates/ Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Concurrent treatment with corticosteroids (or equivalent) except as use for the prophylactic medication regimen, treatment of acute hypersensitivity reactions, or unless chronic treatment (initiated > 6 months prior to study entry) at low dose (<20 mg methyl prednisolone or equivalent)
* Concomitant or with a 4-week period administration of any other experimental drug under investigation
* Concomitant chemotherapy, hormonal therapy, or immunotherapy
* Prior palliative surgery (open and closure, passage operation)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | about 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea